CLINICAL TRIAL: NCT05831982
Title: The Effect of a Complex Person-centered Exercise and Nutrition Intervention for Frail Older Patients on Functional Decline, Quality of Life and Readmissions - A Randomized Controlled Trial.
Brief Title: Exercise and Nutrition Intervention for Frail Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Laurine Nilsson, Physiotherapist, PhD student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-215
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Frailty
Keywords: older; frailty; strength training; nutrition
MeSH Terms: conditions — Frailty | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Due to the vulnerable group masking was not possible for care provider or baseline tester, but randomization will take place after baseline tests have been performed. Tester at 15 and 26 weeks will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (A) (Experimental): Intervention focusing on strength training and nutritional optimization.
  Interventions: Other: Person-centered strength training and nutrition intervention
- Control (B) (Active Comparator): Usual care. Physiotherapy (type of training decided by the physiotherapist) without nutritional intervention.
  Interventions: Other: Standard training

INTERVENTIONS:
Other: Person-centered strength training and nutrition intervention — Focus on high intensity strength training and nutrition intervention with focus on energy and protein intake. Focus on social relations
  Arms: Intervention (A)
Other: Standard training — Training as usual when discharged with a rehabilitation plan.
  Arms: Control (B)

SUMMARY:
The objective of this study is to evaluate the effect of a person-centered training and nutrition intervention six month after discharge in acutely admitted frail old medical patients on physical function. Secondly, to evaluate the effect on frailty, quality of life, health literacy, nutrition, readmissions, death and consumption of home care costs.

DETAILED DESCRIPTION:
Evidence on how to improve physical function and avoid unnecessary readmissions for frail hospitalized older medical patients is not established as yet. In Denmark, the few studies performed have not succeeded in showing a significant difference in physical function or quality of life, due to sector barriers, low compliance and uni-dimensional interventions and none of the studies addressed readmissions and or described a patient-centered approach.

This research project will address this serious individual and societal challenge by testing and evaluating a person-centered complex intervention with emphasis on the patients´ own focus and goals. To increase the probability of developing a successful intervention with the patient in focus we have completed two qualitative studies with patients and health professionals. The primary results from these studies indicate that the pedagogical approach of the involved healthcare professional is important for establishing a good relation. Patients had a desire of being more active, but after four week only a minority had their own expectations fulfilled. Furthermore, the patients expressed that social relations had the potential of increasing adherence to training sessions. Furthermore, a citizen's panel has been established, and possible elements important for the intervention were discussed on behalf of their own experiences with the healthcare system. The results of these qualitative studies and the latest evidence contributed to the development of the current intervention study.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years old
* Acutely admitted with a medical focus at Aalborg University Hospital, South.
* Living in Aalborg Municipality (except 9230 Svenstrup, 9240 Nibe, 9293 Kongerslev, 9381 Sulsted, and 9382 Tylstrup)
* Able to walk (assistance is ok) before admission.
* Speak and understand Danish.

Exclusion Criteria:

* Discharged with rehabilitatinplan for physiotherapy within the last 30 days.
* Dementia or other cognitive impairments.
* Terminal ill.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 26 weeks
  A group of measures that combines the results of the gait speed, chair stand and balance tests

SECONDARY OUTCOMES:
Timed Up and Go | 26 weeks
  A simple test used to assess a person's mobility and requires both static and dynamic balance.
Timed Up and Go | 15 weeks
  A simple test used to assess a person's mobility and requires both static and dynamic balance.
Grip strength | 26 weeks
  Measures the muscular strength or the maximum force generated using a hand held dynamometer
Grip strength | 15 weeks
  Measures the muscular strength or the maximum force generated using a hand held dynamometer
Tilburg Frailty Indicator | 26 weeks
  The Tilburg Frailty Indicator (TFI) is a self-report user-friendly questionnaire for assessing multidimensional frailty among community-dwelling older people
Tilburg Frailty Indicator | 15 weeks
  The Tilburg Frailty Indicator (TFI) is a self-report user-friendly questionnaire for assessing multidimensional frailty among community-dwelling older people
Clinical Frailty Scale (CFS) | 26 weeks
  The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill)
Clinical Frailty Scale (CFS) | 15 weeks
  The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill)
EQ5D-5L | 26 weeks
  A descriptive system which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health)
EQ5D-5L | 15 weeks
  A descriptive system which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health)
Body mass, body fat mass and body muscle mass | 26 weeks
  Inbody270 measurement. I scale measuring mass, fat mass and muscle mass at the same time. Measured in kg.
Body mass, body fat mass and body muscle mass | 15 weeks
  Inbody270 measurement. I scale measuring mass, fat mass and muscle mass at the same time. Measured in kg.
Admission | 26 weeks.
  Number of admissions
Admission | 15 weeks.
  Number of admissions
Home care | 26 weeks.
  Hours of home care
Home care | 15 weeks.
  Hours of home care
Other healthcare services | 26 weeks.
  ex. Occupational therapy or psychologist
Short Physical Performance Battery (SPPB) | 15 weeks
  A group of measures that combines the results of the gait speed, chair stand and balance tests
Height | Baseline
  Measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Laurine Nilsson, PhD stud., Principal Investigator — Aalborg University Hospital; Jane Andreasen, Assoc. prof., Study Chair — Aalborg University Hospital and Aalborg Municipality; Mette Holst, Study Chair — Aalborg University Hospital and Aalborg University; Morten Villumsen, Study Chair — Aarhus Municipality, Denmark
Locations (1):
- Aalborg Municipality, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Rossi PG, Carnavale BF, Farche ACS, Ansai JH, de Andrade LP, Takahashi ACM. Effects of physical exercise on the cognition of older adults with frailty syndrome: A systematic review and meta-analysis of randomized trials. Arch Gerontol Geriatr. 2021 Mar-Apr;93:104322. doi: 10.1016/j.archger.2020.104322. Epub 2020 Dec 10. PMID 33360014
- [Background] Dedeyne L, Deschodt M, Verschueren S, Tournoy J, Gielen E. Effects of multi-domain interventions in (pre)frail elderly on frailty, functional, and cognitive status: a systematic review. Clin Interv Aging. 2017 May 24;12:873-896. doi: 10.2147/CIA.S130794. eCollection 2017. PMID 28579766
- [Background] Andreasen J, Aadahl M, Sorensen EE, Eriksen HH, Lund H, Overvad K. Associations and predictions of readmission or death in acutely admitted older medical patients using self-reported frailty and functional measures. A Danish cohort study. Arch Gerontol Geriatr. 2018 May-Jun;76:65-72. doi: 10.1016/j.archger.2018.01.013. Epub 2018 Feb 13. PMID 29462759
- [Background] Nilsson L, Holst M, Villumsen M, Andreasen J. Maintenance of own health after acute hospitalization - older people's experiences and perspectives on physical activity and nutrition. Physiother Theory Pract. 2024 Jan 2;40(1):100-109. doi: 10.1080/09593985.2022.2122912. Epub 2022 Oct 3. PMID 36189947
- [Background] Rasmussen RL, Holst M, Nielsen L, Villumsen M, Andreasen J. The perspectives of health professionals in Denmark on physical exercise and nutritional interventions for acutely admitted frail older people during and after hospitalisation. Health Soc Care Community. 2020 Nov;28(6):2140-2149. doi: 10.1111/hsc.13025. Epub 2020 Jun 1. PMID 32483900
- [Background] Baert V, Gorus E, Mets T, Geerts C, Bautmans I. Motivators and barriers for physical activity in the oldest old: a systematic review. Ageing Res Rev. 2011 Sep;10(4):464-74. doi: 10.1016/j.arr.2011.04.001. Epub 2011 May 5. PMID 21570493